CLINICAL TRIAL: NCT00777556
Title: Plan B® 1.5 Emergency Contraception Actual Use Study in Adolescents
Brief Title: Emergency Contraception Actual Use Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR-LEV-302
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-09

CONDITIONS: Emergency Contraception
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DR-104 (Experimental): One tablet for emergency contraception
  Interventions: Drug: DR-104

INTERVENTIONS:
Drug: DR-104 — One 1.5 mg tablet of levonorgestrel for emergency contraception within 72 hours following unprotected sexual intercourse.
  Other Names: Plan B® 1.5; Plan B One-Step®; levonorgestrel

SUMMARY:
This is a non-comparative case series study to assess the ability of females 11-16 years of age, inclusive, who are requesting emergency contraception (EC) to use the study product, DR-104 (Plan B® 1.5), appropriately and safely without provider counseling.

DETAILED DESCRIPTION:
To simulate an over-the-counter (OTC) setting, each potential subject was expected to read the label text on the outside of the study package and determine whether and how to use the study product without provider direction or assistance. The study product, Plan B® 1.5, was to be dispensed only to those subjects who appropriately self-selected and indicated that they wanted to participate in the study and receive study product. Subjects could also appropriately self-select not to use the study product.

Follow-up contact was to be conducted at approximately one, four, and eight weeks following the date the subject was dispensed study product. At these contacts, subjects answered questions regarding product use, health problems since last contact, and pregnancy status. Subjects were not to be permitted to enroll more than once in this Actual Use Study, however to assess repeat use of emergency contraceptives (EC) (use in addition to the study product) subjects were also queried at the one-, four-, and eight-week follow-up contacts regarding use of additional EC.

ELIGIBILITY:
Inclusion Criteria:

* Female and 11-16 years of age, inclusive
* Subject must be requesting emergency contraception for her own use (not for use by another person) and for current (not future) use
* Subject can read and understand English, according to her own judgment
* Others as dictated by FDA-approved protocol

Ages: 11 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 343 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Research Protocol Chair, Study Chair — Duramed Research, Inc
Locations (5):
- United States (5):
  - Duramed Research Investigational Site, San Francisco, California
  - Duramed Research Investigational Site, Atlanta, Georgia
  - Duramed Research Investigational Site, Minneapolis, Minnesota
  - Duramed Research Investigational Site, Philadelphia, Pennsylvania
  - Teva Investigational Site, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three hundred and seventy-nine candidates were screened.
Period: Overall Study
Arm/Group | DR-104
Started | 343 (Enrolled; signed informed consent)
Dispensed Product | 307
Safety Population | 299 (Participants who used the product; two were given product in error (inappropriately self-selected))
Used Product | 297
Completed | 277 (Completed all 3 follow-up visits)
Not Completed | 66
Not completed — Inappropriate self-selection | 34
Not completed — Dispensed but did not use product | 12
Not completed — Did not complete all 3 follow-up visits | 20

BASELINE CHARACTERISTICS:
Arm/Group | DR-104
Number analyzed (Participants) | 343
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 343
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Customized [Number; unit: participants]
  11-13 years old | 3
  14 years old | 35
  15 years old | 100
  16 years old | 140
  17 years old | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Latina | 147
  African-American | 48
  Multiracial | 23
  White | 39
  Asian/Pacific Islander | 68
  Native American/Alaskan Native | 1
  Other | 17
Ethnic Latina/Hispanic [Number; unit: participants] — Do you describe yourself as ethnic Latina/Hispanic?
  participants
    No answer | 17
    Yes | 169
    No | 151
    Don't know | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Appropriately Self-selected DR-104 (Plan B® 1.5) When Dispensed Under Simulated Over-the-counter (OTC) Conditions
Description: The percentage of participants who appropriately self-selected Plan B® 1.5 at the Screening/Enrollment Visit after reading the product label. Following the standard norms for a therapy to over-the-counter (Rx-to-OTC) switch process, this outcome is an evaluation of potential consumers' ability to self-diagnose the condition and that treatment with the product is appropriate for them.
Time Frame: Day 1
Population: Enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DR-104
Number analyzed (Participants) | 343
percentage of participants | 90.1 [NA to 86.4] — Not part of analysis plan

2. Primary Outcome: Percentage of Participants Who Correctly Used DR-104 When Dispensed Under Simulated OTC Conditions
Description: The percentage of participants who having appropriately self-selected and been dispensed Plan B® 1.5, correctly used it according to product labeling. Correct use was considered to have occurred if participants reported at the Week 1 follow-up contact that she took Plan B® 1.5 within 72 hours following unprotected sexual intercourse. Following the standard norms for a therapy to over-the-counter (Rx-to-OTC) switch process, this outcome is an evaluation of potential consumers' ability to self-treat with the product according to the product instructions.
Time Frame: Week 1
Population: Eligible participants who appropriately self-selected and used the product.
Measure: Number (95% Confidence Interval); unit: percentage of treated participants
Arm/Group | DR-104
Number analyzed (Participants) | 297
percentage of treated participants | 88.6 [NA to 84.4] — not part of analysis plan

3. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: Treatment-emergent adverse events included adverse events reported during the protocol-specified following up contacts at weeks 1, 4 and 8 or at any other participant contact for participants who took study drug.
Time Frame: Day 1 to week 8
Population: Safety population of participants who took study drug
Measure: Number; unit: participants
Arm/Group | DR-104
Number analyzed (Participants) | 299
participants
  At least one TEAE | 43
  Withdrawn from study due to an AE | 0
  At least one SAE | 1

4. Secondary Outcome: Participants Summarized by Repeat Use of Emergency Contraception (EC)
Description: As each participant dispensed Plan B® 1.5 was only given one tablet, repeat use of emergency contraception (EC) indicates use of an EC product other than the study product. Categories reflect the number of repeat uses.
Time Frame: up to week 8
Population: Participants dispensed the product
Measure: Number; unit: participants
Arm/Group | DR-104
Number analyzed (Participants) | 307
participants
  Repeat uses: 0 | 251
  Repeat uses: 1 | 38
  Repeat uses: 2 | 16
  Repeat uses: 3 | 2

ADVERSE EVENTS:
Time Frame: Day 1 to week 8. Unresolved AEs and pregnancies were followed until resolved.
Description: Includes participants who took study drug. AE information was solicited during scheduled contacts on weeks 1, 4 and 8.
Arm/Group | DR-104
Serious Adverse Events (participants affected / at risk) | 1/299
Other Adverse Events (participants affected / at risk) | 0/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DR-104 (N=299)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.